CLINICAL TRIAL: NCT06186089
Title: Effects of Total Gastrectomy or Double Track Reconstruction on Gut Microbiome and Cognitive Function in Patients With Proximal Gastric Cancer
Brief Title: Effect of Gastrectomy on Gut Microbiome and Cognitive Function
Status: Recruiting | Type: Observational
Sponsor: Jiangjiang Bi (Other)
Responsible Party: Sponsor-Investigator, Jiangjiang Bi, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: JJBi 2023
Record Dates: First submitted 2023-12-07; First posted 2023-12-29 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Perioperative Neurocognitive Disorders; Gastric Cancer
Keywords: Perioperative neurocognitive disorders; proximal gastric cancer; gut microbiota; double-tract reconstruction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faeces and Peripheral Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Probiotics (PR): Patients undergoing total gastrectomy take probiotics qd for 3 months after surgery.
  Interventions: Dietary Supplement: probiotics
- Total gastrectomy (TG): Patients undergoing total gastrectomy
- Double-tract reconstruction (DTR): Patients undergoing double-tract reconstruction

INTERVENTIONS:
Dietary Supplement: probiotics — patients undergoing total gastrectomy take probiotics qd for 3 months
  Groups: Probiotics (PR)

SUMMARY:
Perioperative neurocognitive disorders is a common postoperative complication in elderly surgical patients. The role of gut microbiota in cognitive function has been concerned in recent years. Studies suggests that gastrointestinal surgery may affect the gut microbiota, and the effect varies between surgical procedures. In this study, the investigators will compare the differences of gut microbiota between total gastrectomy and double-tract reconstruction, to investigate the effect of gastric acid on the gut microbiota colonizing, and the effect of different surgical procedures on the postoperative cognitive function of proximal gastric cancer patients.

DETAILED DESCRIPTION:
Perioperative neurocognitive disorders is a common postoperative complication in elderly surgical patients, especially in gastrointestinal tumors and cardiac on-pump surgery, and the mechanism is not clear yet. The role of gut microbiota in cognitive function has been concerned in recent years, and the applicant's previous study also found significant differences in the composition of gut microbiota and metabolites in elderly orthopedic surgical patients with postoperative cognitive dysfunction compared with the control group, and that the differential metabolites were mainly enriched in the metabolic pathway of protein digestion and absorption. Studies suggests that gastrointestinal surgery may affect the gut microbiota, and the effect varies between surgical procedures. The incidence of proximal gastric cancer is increasing. In order to prevent severe gastroesophageal reflux, total gastrectomy is mostly performed. However, after total gastrectomy, food directly enters into the intestine, followed by insufficient mixing of gastric acid and food. Patients are prone to nutrient absorption disorders, which may cause changes in gut microbiota. The double-tract reconstruction allows food to enter the distal gastrointestinal tract via two pathways, successfully solving the problems of gastroesophageal reflux, gastroparesis, and long-term nutritional disorders in patients after proximal gastrectomy. In this study, the investigators aim to investigate the effect of gastric acid on the gut microbiota colonizing, and the effect of different surgical procedures on the postoperative cognitive function of proximal gastric cancer patients. The investigators will compare the differences of gut microbiota between total gastrectomy and double-tract reconstruction by 16S ribosomal ribonucleic acid (rRNA) gene sequencing and metabonomics technology, and evaluate the postoperative cognitive function by Mini-mental State Examination scales and Montreal Cognitive Assessment scales.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of proximal gastric cancer and will be performed gastrectomy
2. American Society of Anesthesiologists (ASA) classification I-III
3. Aged 40-80 years
4. Perioperative consciousness

Exclusion Criteria:

1. Central nervous system and psychological disorders
2. Chronic use of sedatives, antidepressants within the last year
3. Parkinson's disease
4. Severe immunosuppression
5. Severe hearing or vision impairment
6. Drug dependence; alcoholism
7. Inability to communicate with a physician

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing proximal gastric cancer surgery with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 1 day before surgery; 1 day, 7 days, 3 months and 12 months after surgery
  The participants will be evaluated by Mini-mental State Examination scales, and diagnosed as cognitive dysfunction if score < 24.
Cognitive function | 1 day before surgery; 1 day, 7 days, 3 months and 12 months after surgery
  The participants will be evaluated by Montreal Cognitive Assessment scales, diagnosed as cognitive dysfunction if score < 26
Composition and diversity of gut microbiota | 1 day before surgery and 7 days after surgery
  It will be tested by 16s rRNA gene sequencing.

SECONDARY OUTCOMES:
Inflammatory factor | preoperation, 30 minutes and 24 hours after surgery
  Interleukin-1β (IL-1β), IL-6, tumor necrosis factor-α (TNF-α), C reactive protein (CRP) will be tested by ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangjiang Bi, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the Nomenclature of Cognitive Change Associated with Anaesthesia and Surgery-2018. Anesthesiology. 2018 Nov;129(5):872-879. doi: 10.1097/ALN.0000000000002334. PMID 30325806
- [Background] Naseer MI, Bibi F, Alqahtani MH, Chaudhary AG, Azhar EI, Kamal MA, Yasir M. Role of gut microbiota in obesity, type 2 diabetes and Alzheimer's disease. CNS Neurol Disord Drug Targets. 2014 Mar;13(2):305-11. doi: 10.2174/18715273113126660147. PMID 24059313
- [Background] Mulak A, Bonaz B. Brain-gut-microbiota axis in Parkinson's disease. World J Gastroenterol. 2015 Oct 7;21(37):10609-20. doi: 10.3748/wjg.v21.i37.10609. PMID 26457021
- [Background] Bi J, Xu Y, Li S, Zhan G, Hua D, Tan J, Chi X, Xiang H, Guo F, Luo A. Contribution of preoperative gut microbiota in postoperative neurocognitive dysfunction in elderly patients undergoing orthopedic surgery. Front Aging Neurosci. 2023 Feb 17;15:1108205. doi: 10.3389/fnagi.2023.1108205. eCollection 2023. PMID 36875700
- [Background] Zhan G, Yang N, Li S, Huang N, Fang X, Zhang J, Zhu B, Yang L, Yang C, Luo A. Abnormal gut microbiota composition contributes to cognitive dysfunction in SAMP8 mice. Aging (Albany NY). 2018 Jun 10;10(6):1257-1267. doi: 10.18632/aging.101464. PMID 29886457
- [Background] Maksimaityte V, Bausys A, Kryzauskas M, Luksta M, Stundiene I, Bickaite K, Bausys B, Poskus T, Bausys R, Strupas K. Gastrectomy impact on the gut microbiome in patients with gastric cancer: A comprehensive review. World J Gastrointest Surg. 2021 Jul 27;13(7):678-688. doi: 10.4240/wjgs.v13.i7.678. PMID 34354801
- [Background] Jahansouz C, Staley C, Bernlohr DA, Sadowsky MJ, Khoruts A, Ikramuddin S. Sleeve gastrectomy drives persistent shifts in the gut microbiome. Surg Obes Relat Dis. 2017 Jun;13(6):916-924. doi: 10.1016/j.soard.2017.01.003. Epub 2017 Jan 4. PMID 28279578
- [Background] Erawijantari PP, Mizutani S, Shiroma H, Shiba S, Nakajima T, Sakamoto T, Saito Y, Fukuda S, Yachida S, Yamada T. Influence of gastrectomy for gastric cancer treatment on faecal microbiome and metabolome profiles. Gut. 2020 Aug;69(8):1404-1415. doi: 10.1136/gutjnl-2019-319188. Epub 2020 Jan 16. PMID 31953253
- [Background] Cavin JB, Couvelard A, Lebtahi R, Ducroc R, Arapis K, Voitellier E, Cluzeaud F, Gillard L, Hourseau M, Mikail N, Ribeiro-Parenti L, Kapel N, Marmuse JP, Bado A, Le Gall M. Differences in Alimentary Glucose Absorption and Intestinal Disposal of Blood Glucose After Roux-en-Y Gastric Bypass vs Sleeve Gastrectomy. Gastroenterology. 2016 Feb;150(2):454-64.e9. doi: 10.1053/j.gastro.2015.10.009. Epub 2015 Oct 23. PMID 26481855
- [Background] Bianchi VE, Herrera PF, Laura R. Effect of nutrition on neurodegenerative diseases. A systematic review. Nutr Neurosci. 2021 Oct;24(10):810-834. doi: 10.1080/1028415X.2019.1681088. Epub 2019 Nov 4. PMID 31684843
- [Background] van de Wouw M, Boehme M, Lyte JM, Wiley N, Strain C, O'Sullivan O, Clarke G, Stanton C, Dinan TG, Cryan JF. Short-chain fatty acids: microbial metabolites that alleviate stress-induced brain-gut axis alterations. J Physiol. 2018 Oct;596(20):4923-4944. doi: 10.1113/JP276431. Epub 2018 Aug 28. PMID 30066368
- [Background] Martin CR, Osadchiy V, Kalani A, Mayer EA. The Brain-Gut-Microbiome Axis. Cell Mol Gastroenterol Hepatol. 2018 Apr 12;6(2):133-148. doi: 10.1016/j.jcmgh.2018.04.003. eCollection 2018. PMID 30023410